CLINICAL TRIAL: NCT02968264
Title: Tetralogy of Fallot for Life
Acronym: TOF-LIFE
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Other Study IDs: TOF-LIFE 2.0 2015-06-11
Record Dates: First submitted 2016-01-04; First posted 2016-11-18 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Tetralogy of Fallot; Congenital Heart Disease; Congenital Heart Defect
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TOF participants: Tetralogy of fallot patients at any age

SUMMARY:
The aim is to conduct a prospective multi-centre international inception cohort study with an enrollment goal of 3,000 TOF patients and 2 year follow-up post-repair. The proposed sample size and methodology will result in statistically powerful results to allow for evidence-based change to current TOF surgical practices.

DETAILED DESCRIPTION:
Background: Tetralogy of Fallot (TOF) is the most common cyanotic heart defect consisting of 7-10% of all congenital heart disease with an estimated annual global incidence rate of 38,000. It is fatal if untreated; only 50% of patients are alive at 1 year of age. Surgery has dramatically improved the survival so that >95% of repaired TOF children are alive by one year. The initial justified enthusiasm for the benefit of surgical therapy are now tempered by the findings of late sudden cardiac death secondary to right ventricular (RV) dysfunction. The original trans-ventricular/trans-annular patching repair results in significant pulmonary insufficiency which leads to RV dilation, subsequent functional tricuspid regurgitation, atrial arrhythmias, and eventual RV failure and ventricular arrhythmias. In attempt to break this cycle, an increasing number of patients are undergoing late pulmonary valve implantation.

Recognizing that the RV adapts to stress signals has led to the idea that leaving mixed residual stenosis and regurgitation may yield to an adaptive change that limits RV dilation while still allowing for adequate cardiac output. Early attempts to limit pulmonary insufficiency and RV damage involve minimal trans-annular patching or complete annulus preservation (AP). Emerging data suggest that patients with a mixed lesion have improved survival, so that 96.6% are alive at 25-years in comparison to 85-90% survival for the conventional technique.

Preliminary Data: A review of data comparing AP to TAP repair at our institution (n=185, AP repair=124, TAP=61) demonstrated that at 10-15 year follow-up those who received an AP repair had smaller RV volumes and pulmonary regurgitant jet width. They were also seen to have improved exercise capacity as measure by VO2 max tests. The AP technique also has been seen to significantly decrease the risk of reoperation in comparison to TAP, 11% and 29% respectively.

Current Problem: Although trans-ventricular VSD closure along with a TAP is known to result in increased risk of long-term morbidity and mortality, it continues to be the predominant repair strategy implemented globally according to STS/EACTS databases. Reasons for this are:

* Trans-ventricular/TAP approach is technically easier than annulus preservation, which often requires multiple pump runs
* There is a fear of leaving too much obstruction
* High quality evidence supporting one approach over the other is lacking.

Gaps in Literature

1. Most data on the impact of surgical strategy emerge from single centre experiences that are retrospective and based on small patient population. This makes the results difficult to standardize to the general TOF population.
2. Retrospective registry data published by STS and EACTS omit many crucial surgical and clinical variables that can potentially impact outcomes.
3. None of the current evidence are based on anatomically matched/adjusted patients

ELIGIBILITY:
Inclusion Criteria:

* TOF with RVOT stenosis. TOF is defined as anterio-cephalad deviation of the ventricular outlet septum with no more than 50% aortic override and a single outflow VSD.
* TOF with pulmonary atresia and confluent pulmonary arteries.
* Admitted with intent to treat (i.e. patient planned to undergo a primary or staged repair).
* Patients with coronary artery anomalies, right aortic arch, and 22q11 deletion may be included

Exclusion Criteria:

* TOF with absent pulmonary valve
* Other major cardiac anomalies such as AVSD, multiple VSDs, right atrial isomerism, and MAPCAs. In this instance, the definition of MAPCAs does not include dilated bronchial collateral arteries.
* Unbalanced ventricles precluding biventricular repair
* Major genetic abnormalities/syndromes e.g. trisomy 13,18, and 21
* Major extra cardiac anomalies e.g. diaphragmatic hernia, omphalocele, absent sternum, cerebral palsy
* Infective endocarditis as an indication for intra-cardiac repair
* Stroke in the last 30 days prior to palliation or intra-cardiac repair
* Known diagnosis of HIV or hepatitis B
* Any previous cardiac procedures
* Patient's circumstance that precludes completion of follow-up telephone call and/or obtaining information from the 2-year cardiology follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TOF patients of any age undergoing their first cardiac intervention. Please refer to the eligibility criteria for more details.
Sampling Method: Non-Probability Sample
Enrollment: 1108 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
RV physiology and morphology | 2 years post-repair
  To determine the association between baseline morphology, surgical repair technique (various surgical strategies for VSD closure and managing the RVOT), and RV physiology and morphology at 2 years obtained from echocardiogram studies.

SECONDARY OUTCOMES:
Number of patients undergoing various palliation procedures and surgical repair strategies | 2 years
  To determine the pattern of palliation procedures (BT shunt, RVOT stent, or balloon dilation), surgical repair strategy (staged versus primary repair), and surgical repair technique (AP, minimal TAP, standard TAP) at participating centres.
Cardiovascular mortality rate | 30 days and 2 years after repair
  To determine the 30-day and 2 year cardiovascular mortality rate (for equivalent patients) after primary and staged repair.
Rate of palliation failure | 2 years
  To determine the rate of palliation failure following various palliation techniques
Effect of palliation procedures on cardiac morphology | 2 years
  To determine the possible effect of palliative procedures (BT shunts, balloon dilation, stent insertion) on cardiac morphology (growth of the infundibular chamber, the pulmonary annulus and PA branches' diameter) and subsequent repair technique.
Post-operative restrictive physiology | 2 years
  To determine the relationship between repair technique/strategy and prevalence of postoperative restrictive physiology as defined by the presence of antegrade flow in pulmonary artery during atrial contraction on echocardiogram.
Cardiac re-interventions | 2 years
  To determine the relationship between TOF repair strategy/technique on the incidence and prevalence of cardiac re-interventions (e.g. pulmonary valve implantation, RVOT stent insertion or balloon dilatation)
RV physiology and morphology following TOF pulmonary atresia repair | 2 years
  To determine the right ventricular morphological and physiological adaptations to severe pulmonary stenosis or regurgitation using repaired TOF pulmonary atresia as a model. For example RV/LV end diastolic and systolic diameter ratio. RV and LV wall thickness relation to outflow gradient obtained by echocardiogram studies.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Van Arsdell, MD, Principal Investigator — University of California, Los Angeles; Richard Whitlock, MD, PhD, Principal Investigator — Population Health Research Institute
Locations (20):
- United States (2):
  - Nemours Children's Hospital, Orlando, Florida
  - Morgan Stanley Children's Hospital, New York, New York
- Royal Children's Hospital, Parkville, Victoria, Australia
- Hospital for Sick Children, Toronto, Ontario, Canada
- China (6):
  - West China Hospital, Chengdu, Sichuan
  - Beijing Fuwai Hospital, Beijing
  - Guangzhou Women and Children's Medical Center, Guangdong
  - Guangdong Cardiovascular Institute, Guangdong
  - Shanghai Children's Medical Centre, Shanghai
  - Shanghai Xinhua Hospital, Shanghai
- India (2):
  - Fortis Escorts Heart Institute, New Delhi, National Capital Territory of Delhi
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institutev, Mumbai
- National Cardiovascular Center Harapan Kita, Jakarta, Indonesia
- Okayama University Hospital, Okayama, Japan
- Manmohan Cardiothoracic Vascular and Transplant Center, Kathmandu, Nepal
- Academician E.N. Meshalkin Research, Novosibirsk, Russia
- Saudi Arabia (2):
  - King Abdulaziz University Hospital, Jeddah, Mecca Region
  - King Faisal Specialist Hospital and Research Centre - Jeddah, Jeddah
- Asan Medical Center, Seoul, South Korea
- Children's Cardiac Center - Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarris GE, Comas JV, Tobota Z, Maruszewski B. Results of reparative surgery for tetralogy of Fallot: data from the European Association for Cardio-Thoracic Surgery Congenital Database. Eur J Cardiothorac Surg. 2012 Nov;42(5):766-74; discussion 774. doi: 10.1093/ejcts/ezs478. PMID 23087090
- [Background] Al Habib HF, Jacobs JP, Mavroudis C, Tchervenkov CI, O'Brien SM, Mohammadi S, Jacobs ML. Contemporary patterns of management of tetralogy of Fallot: data from the Society of Thoracic Surgeons Database. Ann Thorac Surg. 2010 Sep;90(3):813-9; discussion 819-20. doi: 10.1016/j.athoracsur.2010.03.110. PMID 20732501
- [Background] Gatzoulis MA, Balaji S, Webber SA, Siu SC, Hokanson JS, Poile C, Rosenthal M, Nakazawa M, Moller JH, Gillette PC, Webb GD, Redington AN. Risk factors for arrhythmia and sudden cardiac death late after repair of tetralogy of Fallot: a multicentre study. Lancet. 2000 Sep 16;356(9234):975-81. doi: 10.1016/S0140-6736(00)02714-8. PMID 11041398
- [Background] d'Udekem Y, Galati JC, Rolley GJ, Konstantinov IE, Weintraub RG, Grigg L, Ramsay JM, Wheaton GR, Hope S, Cheung MH, Brizard CP. Low risk of pulmonary valve implantation after a policy of transatrial repair of tetralogy of Fallot delayed beyond the neonatal period: the Melbourne experience over 25 years. J Am Coll Cardiol. 2014 Feb 18;63(6):563-8. doi: 10.1016/j.jacc.2013.10.011. Epub 2013 Oct 30. PMID 24513776
- [Background] Pondorfer P YT, Cheung M, Ashburn D, Manlhiot C, McCrindle B, Mertens L, Grosse-Wortmann L, Redington A, Van Arsdell G. Abstract 18833: Annulus Preservation Strategy Improves Late Outcomes in Tetralogy of Fallot: An Anatomical Equivalency Study. Circulation. 2014;130:A18833.